CLINICAL TRIAL: NCT02723656
Title: Using Cancer Registry Data to Promote Proactive Tobacco Cessation Among Adult Cancer Survivors U48
Brief Title: Proactive Care Coordination for Cancer Survivors Who Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-01069
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cancer
Keywords: smoking; cancer; cancer registry; smoking cessation
MeSH Terms: conditions — Neoplasms; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proactive mailed care coordination (Active Comparator)
  Interventions: Behavioral: Online Referral NYS Quitline
- Proactive telephone care coordination. (Active Comparator)
  Interventions: Behavioral: Tobacco cessation counseling and coordination of cessation medications

INTERVENTIONS:
Behavioral: Online Referral NYS Quitline — Care coordinator will make an online referral to the NYS Quitline.
  Arms: Proactive mailed care coordination
Behavioral: Tobacco cessation counseling and coordination of cessation medications — Care coordinator will obtain verbal consent to transfer the patient to the NYS Quitline via 3-way call (warm transfer). The care coordinator will also assist the patient in obtaining NRT from a regular care provider, then call the patient every three months for 12 months to assess current smoking and offer to help smokers obtain additional cessation counseling and medications.
  Arms: Proactive telephone care coordination.

SUMMARY:
This is a population-based randomized controlled trial of 600 patients with a diagnosis of cancer in the past 2 years and registry indicating smoking at the time of diagnosis, that will inform critical questions regarding the relative efficacy of care coordination options, the reliability of Electronic Health Record (EHR) tobacco use data, and how patients will react to proactive tobacco related communications. Investigators will compare the reach and efficacy of two proactive approaches to enrolling cancer survivors in tobacco treatment (Arm 1: mailed care coordination vs. Arm 2: telephone care coordination) using a two-arm randomized design at two urban cancer centers, and will explore cancer survivor attitudes and preferences about proactive tobacco treatment.

ELIGIBILITY:
Inclusion Criteria:

* ICD 9 cancer diagnosis seen at each site in the past two years
* Documentation of current smoking in the cancer registry.

Exclusion Criteria:

* Dementia
* Stage IV or Stage IIIB cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in the study's original proactive outreach cohort of N=600 who complete at least one call with the Quitline | 12 Months

SECONDARY OUTCOMES:
biochemically validated 7-day abstinence | 6 Months, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krebs, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States